CLINICAL TRIAL: NCT02754674
Title: Comparison of Femoral Tunnel Placement, Geometry and Clinical Outcome Using Two Anterior Cruciate Ligament Reconstruction Technique; Transportal Technique and Outside in Technique With Remnant Preservation. Prospective Randomized Trial
Brief Title: Comparison of Femoral Tunnel and Clinical Outcome Using Two Anterior Cruciate Ligament Reconstruction Techniques
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SMC2013-07-097-001
Record Dates: First submitted 2015-02-22; First posted 2016-04-28 (Estimated); Results first posted 2019-12-20 (Actual); Last update posted 2019-12-20 (Actual); Status verified 2017-12

CONDITIONS: Rupture of Anterior Cruciate Ligament
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Transportal (Experimental): this is a type of anterior cruciate ligament reconstruction. this arm for patients who underwent operation with transportal technique
  Interventions: Procedure: type of anterior cruciate ligament reconstruction
- Outside in (Experimental): this is a type of anterior cruciate ligament reconstruction. this arm for patients who underwent operation with patients who underwent operation with outside in technique
  Interventions: Procedure: type of anterior cruciate ligament reconstruction

INTERVENTIONS:
Procedure: type of anterior cruciate ligament reconstruction — comparison of different types of anterior cruciate ligament reconstruction. transportal technique is double bundle graft using flexible reamer, outside-in technique is single bundle graft with remnant preservation

SUMMARY:
1. Purpose :To compare of femoral tunnel placement, tunnel geometry and clinical outcome using two anterior cruciate ligament reconstruction techniques ; transportal technique with flexible reamer and single bundle outside in technique with remnant preservation.
2. Subjects: anterior cruciate ligament (ACL) injury 66 patients

   * Double bundle transportal technique with flexible reamer: 33
   * Single bundle outside in technique with remnant preservation: 33

DETAILED DESCRIPTION:
Anterior cruciate ligament (ACL) injury patients : Total 66

1. Double bundle transportal technique with flexible reamer: 33

   * Advantage: more normal ACL reconstruction than single bundle technique
   * Disadvantage: to make the two bone tunnel must remove all the residual tissue.
2. Single bundle outside in technique with remnant preservation: 33

   * Advantage: good for being synovium and revascularization. Remained proprioception function helps to functional recovery.
   * Disadvantage: difficult to ensure of visibility and tunnel drilling in the correct position because of remnant tissue.

ELIGIBILITY:
Inclusion Criteria:

1. Lachman test grade II,III and Pivot shift test grade II,III in physical examination
2. ACL rupture in MRI
3. Age 20~60
4. within 6 months after trauma

Exclusion Criteria:

1. osteoarthritis (OA) change in X-ray
2. History of other ligament injury or ACL reconstruction in uninjured knee.
3. operation history of either ipsilateral or contralateral knee(fracture, etc)

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 67 (Actual)
Dates: Start 2014-05 (Actual); Primary Completion 2014-05 (Actual); Study Completion 2017-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joon Ho Wang, MD, Ph D, Study Chair — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No
if yes, age, sex, physical examination, trauma date, MRI.

REFERENCES:
- [Derived] Wang JH, Lee ES, Lee BH. Paradoxical tunnel enlargement after ACL reconstruction with hamstring autografts when using beta-TCP containing interference screws for tibial aperture fixation- prospectively comparative study. BMC Musculoskelet Disord. 2017 Sep 16;18(1):398. doi: 10.1186/s12891-017-1757-0. PMID 28915914

RESULTS

PARTICIPANT FLOW:
Groups:
- Transportal: this is a type of anterior cruciate ligament reconstruction. this arm for patients who underwent operation with transportal technique
  type of anterior cruciate ligament reconstruction: comparison of different types of anterior cruciate ligament reconstruction.
  transportal technique is double bundle graft using flexible reamer, outside-in technique is single bundle graft with remnant preservation.
- Outside in: this is a type of anterior cruciate ligament reconstruction. this arm for patients who underwent operation with patients who underwent operation with outside in technique
  type of anterior cruciate ligament reconstruction: comparison of different types of anterior cruciate ligament reconstruction.
  transportal technique is double bundle graft using flexible reamer, outside-in technique is single bundle graft with remnant preservation.
Period: Overall Study
Arm/Group | Transportal | Outside in
Started | 34 | 33
Completed | 28 | 26
Not Completed | 6 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Transportal | Outside in | Total
Number analyzed (Participants) | 34 | 33 | 67
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 34 | 33 | 67
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: year] | 29.5 (8) | 33.5 (9.3) | 31.4 (8.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 6 | 12
  Male | 28 | 27 | 55
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  South Korea | 34 | 33 | 67
Time from injury to ACLR [Mean (Standard Deviation); unit: month] | 1.4 (1.6) | 1.5 (1.7) | 1.4 (1.6)
Auto-Graft [Count of Participants; unit: Participants] | 8 | 10 | 18
BMI [Mean (Standard Deviation); unit: kg/m2] | 25.8 (4) | 25.1 (2.9) | 25.5 (3.5)

OUTCOME MEASURES:

1. Primary Outcome: Vascularity of Graft Tendon
Description: For evaluation of graft vascularity, quantitative parameter of area under the curve (AUC) was measured from DCE-MRI by using an image-processing software (IntelliSpace Portal, version 5.0; Philips Healthcare). A musculoskeletal radiologist manually drew the ROIs for intra-articular portion of the ACL graft including synovial membrane at the proximal, middle and distal zones. The software automatically generated time to signal intensity curves and then calculated the quantitative parameter, area under the time to signal intensity curve values, which were acquired by integrating the area under the time to signal intensity curve. To normalize the AUC (nAUC), we divided the AUC of medial gastrocnemius muscle into that of the ACL graft.
Time Frame: 1yr after surgery
Measure: Mean (Standard Deviation); unit: ratio of AUC
Arm/Group | Transportal | Outside in
Number analyzed (Participants) | 28 | 26
ratio of AUC | 2.5 (2.0) | 4.1 (2.5)
Statistical Analysis 1: Comparison: Transportal vs Outside in; Test type: Superiority; p = 0.008, t-test, 2 sided

2. Secondary Outcome: Arthroscopy Grading
Description: Graft continuity was graded as no tears, superficial tear (fibrillation or tear of superficial fibers), or substantial tear (rupture of 1 or more strands).
  Graft tension was graded as taut, mild lax, and lax by probing at knee flexion and extension.
  Synovial coverage of the grafts was graded as excellent (synovial coverage > 80% around graft), fair (coverage > 50%), or poor (coverage < 50%) On the second-look arthroscopic examination, graft continuity, graft tension, graft synovialization, and the presence of cyclops lesions were assessed by a senior surgeon.
Time Frame: 1yr after surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Transportal | Outside in
Number analyzed (Participants) | 21 | 20
Participants
  synovialization: Excellent | 6 | 11
  synovialization: Fair | 9 | 7
  synovialization: Poor | 6 | 2
  continuity: Excellent | 15 | 11
  continuity: Fair | 3 | 8
  continuity: Poor | 3 | 1
  tension: Excellent | 17 | 18
  tension: Fair | 3 | 1
  tension: Poor | 1 | 1
Statistical Analysis 1: Comparison: Transportal vs Outside in; Test type: Superiority; p > 0.05, Chi-squared

3. Secondary Outcome: Clinical Knee Scoring
Description: Lysholm score (ragne 0-100), HSS (hospital for special surgery) score (0-100) , IKDC (international knee doucomentation commitee) subjective score (0-100), Tegner activity scale (0-10).
  All of scores demonstrated that higher score means a better outcomes.
Time Frame: 2 yr after surgery
Measure: Mean (Standard Deviation); unit: score
Arm/Group | Transportal | Outside in
Number analyzed (Participants) | 28 | 26
score
  Lysholm score | 89.1 (8.4) | 90.1 (9.1)
  HSS score | 97.4 (4.0) | 98.7 (3.3)
  IDKC score | 83.6 (9.7) | 87.9 (7.7)
  tegner | 6 (2) | 6 (2)
Statistical Analysis 1: Comparison: Transportal vs Outside in; We used the Kolmogorov-Smirnov test to assess the normality of the data distribution. Student's t-test or the Mann-Whitney U-test was used to analyze intergroup differences. The paired t-test or Wilcoxon signed rank test was used to analyze differences between pre- and postoperative values. Pearson's Chi-square test or Fisher's exact test was used to analyze categorical variables between groups. The statistical significance level was set at .05; Test type: Superiority — Student's t-test or the Mann-Whitney U-test was used to analyze intergroup differences. The paired t-test or Wilcoxon signed rank test was used to analyze differences between pre- and postoperative values. The statistical significance level was set at .05; p > 0.05, t-test, 2 sided

4. Secondary Outcome: Instability
Description: The side-to-side difference was measured using a KT-200- arthrometer (MEDmetric) at 30 lb in 30° of knee flexion.
Time Frame: 2 yr after surgery
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Transportal | Outside in
Number analyzed (Participants) | 28 | 26
mm | 2.6 (1.3) | 1.9 (1.0)
Statistical Analysis 1: Comparison: Transportal vs Outside in; Test type: Superiority; p > 0.05, t-test, 2 sided

5. Secondary Outcome: Graft Maturity (SNQ)
Time Frame: 1 yr after surgery
Measure: Mean (Standard Deviation); unit: SNQ
Arm/Group | Transportal | Outside in
Number analyzed (Participants) | 28 | 26
SNQ | 69.4 (34.7) | 53.1 (24.5)
Statistical Analysis 1: Comparison: Transportal vs Outside in; Test type: Superiority; p = 0.054, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: between 6months and 1 year
Arm/Group | Transportal | Outside in
All-Cause Mortality (participants affected / at risk) | 0/28 | 0/26
Serious Adverse Events (participants affected / at risk) | 0/28 | 0/26
Other Adverse Events (participants affected / at risk) | 0/28 | 0/26
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Transportal (N=28) | Outside in (N=26)
infection (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) — surgical site infection

LIMITATIONS AND CAVEATS:
Technical problems with measurement leading to unreliable or uninterpretable data

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No